CLINICAL TRIAL: NCT01416506
Title: Community-Acquired Pneumonia (CAP) Mycoplasma Surveillance
Brief Title: Community-Acquired Pneumonia (CAP) Surveillance
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15465; NN1010CN (Other: Company Internal)
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Pneumonia
Keywords: Pneumonia, surveillance
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: No Drug

INTERVENTIONS:
Other: No Drug — It's a surveillance

SUMMARY:
Prospective, non-interventional, multi-center study. 7 investigative centers will involved in China. Around 560 CAP outpatients or inpatients will be screened until 56 M. pneumoniae isolates collected.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adult (male or female) ≥18 years old
* Outpatients or inpatients who suffer from CAP

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adult (male or female) >/= 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
In vitro Minimal Inhibitory Concentration Detection | Up to 27 months

SECONDARY OUTCOMES:
In vitro Gene Mutation Detection | Up to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China